CLINICAL TRIAL: NCT02461381
Title: Bayesian Estimation of Diagnostic Performance of Short-term Heart Rate Variability for Diabetic Cardiovascular Autonomic Neuropathy in the Absence of a Gold Standard
Brief Title: Bayesian Estimation of Diagnostic Performance of Diabetic Cardiovascular Autonomic Neuropathy Without a Gold Standard
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Zihui Tang, M.D and Ph.D, Shanghai Tongji Hospital, Tongji University School of Medicine
Other Study IDs: DCANHRVB_Dr.Tang
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Cardiovascular Autonomic Neuropathy (DCAN)
Keywords: Bayesian estimation, short-term heart rate variability, diabetic cardiovascular autonomic neuropathy, diagnostic performance; Diagnostic performance; short-term heart rate variability; diabetic cardiovascular autonomic neuropathy; DCAN

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dr.Tang's research group: This group included diabetic participants with completed both the short-term HRV test and Ewing's test.
  Interventions: Other: not intervention

INTERVENTIONS:
Other: not intervention — This is a cross-sectional study for estimation of diagnostic performance.
  Other Names: nothing

SUMMARY:
This study aimed to estimate sensitivities and specificities of diabetic cardiovascular autonomic neuropathy (DCAN) diagnostic tests using the Bayesian approach without a gold standard in another independence dataset.The reference the values for the short-term HRV were calculated in the investigators' previous study (including 371 healthy subjects). This study dataset contained 200 diabetic patients who completed both the short-term HRV test and Ewing's test. Simultaneous inferences about the population prevalence and the performance of each diagnostic test were possible using the Bayesian approach without a gold standard.

DETAILED DESCRIPTION:
The CAN prevalence is rapidly growing in all populations worldwide. No document has been reported diagnostic performance of short-term heart rate variability (HRV) for diabetic cardiovascular autonomic neuropathy (DCAN) in the Chinese population. This study aimed to estimate sensitivities and specificities of DCAN diagnostic tests using the Bayesian approach, in the absence of a gold standard in another independence dataset.The reference the values for the short-term HRV were calculated in the investigators' previous study (including 371 healthy subjects). This study dataset contained 200 subjects who completed both the short-term HRV test and Ewing's test. Simultaneous inferences about the population prevalence and the performance of each diagnostic test were possible using the Bayesian approach without a gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Survey diabetic participants with undiagnosed CAN, aged 30-90 years, were included in this study.

Exclusion Criteria:

* Some subjects were excluded from the study to eliminate potential confounding factors that may have influenced their CA function. Briefly, the exclusion criteria were as follows:

  1. history or findings of arrhythmia, and hyperthyroidism or hypothyroidism;
  2. pregnancy or lactation; and/or
  3. serious hepatic or renal dysfunctions.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with inclusion and exclusion criteria were recruited from healthy examination centres to assess cardiovascular autonomic function using both the short-term heart rate variability and Ewing's tests.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Diabetic cardiovascular autonomic function evaluate by short-term heart rate variability test | participants will be measured for the duration of outpatient stay, an expected average of two days
  Both short-term heart rate variability and Ewing's test measure diabetic cardiovascular autonomic function
Diabetic cardiovascular autonomic function evaluate by Ewing's test | participants will be measured for the duration of outpatient stay, an expected average of two days
  Both short-term heart rate variability and Ewing's test measure cardiovascular autonomic function

CONTACTS AND LOCATIONS:
Overall Officials: Zihui Tang, M.D and Ph.D, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li Z, Tang ZH, Zeng F, Zhou L. Associations between the severity of metabolic syndrome and cardiovascular autonomic function in a Chinese population. J Endocrinol Invest. 2013 Dec;36(11):993-9. doi: 10.3275/9005. Epub 2013 Jun 17. PMID 23770583
- [Result] Tang ZH, Zeng F, Yu X, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on baroreflex sensitivity in the absence of a gold standard. Int J Cardiol. 2014 Feb 15;171(3):e78-80. doi: 10.1016/j.ijcard.2013.11.100. Epub 2013 Dec 6. No abstract available. PMID 24360155
- [Result] Zeng F, Tang ZH, Li Z, Yu X, Zhou L. Normative reference of short-term heart rate variability and estimation of cardiovascular autonomic neuropathy prevalence in Chinese people. J Endocrinol Invest. 2014 Apr;37(4):385-91. doi: 10.1007/s40618-013-0047-4. Epub 2014 Jan 9. PMID 24633734
- [Result] Tang ZH, Wang L, Zeng F, Li Z, Yu X, Zhang K, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on short-term heart rate variability without a gold standard. BMJ Open. 2014 Oct 6;4(9):e005096. doi: 10.1136/bmjopen-2014-005096. PMID 25287103
- [Result] Tang ZH, Liu J, Zeng F, Li Z, Yu X, Zhou L. Comparison of prediction model for cardiovascular autonomic dysfunction using artificial neural network and logistic regression analysis. PLoS One. 2013 Aug 5;8(8):e70571. doi: 10.1371/journal.pone.0070571. Print 2013. PMID 23940593
- [Derived] Chen J, Yang SB, Liu J, Tang ZH. Diagnostic performance analysis for diabetic cardiovascular autonomic neuropathy based on short-term heart rate variability using Bayesian methods: preliminary analysis. Diabetol Metab Syndr. 2015 Sep 10;7:74. doi: 10.1186/s13098-015-0070-z. eCollection 2015. PMID 26366204